CLINICAL TRIAL: NCT04762264
Title: A 3D Regenerative Scaffold for Inguinal Hernia Repair. MR Imaging and Histological Cross Evidence.
Brief Title: MR Imaging of the 3D Inguinal Hernia Scaffold ProFlor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Giuseppe Amato, Consultant Professor, University of Cagliari
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: MR imaging of ProFlor
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2021-02

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Short term post inguinal hernia repair with ProFlor (Active Comparator): MRI of the pelvic area in patients who underwent inguinal hernia repair with ProFlor from 1 to 3 months before to assess tissue incorporation into the 3D scaffold
  Interventions: Device: ProFlor inguinal hernia device
- Mid term post inguinal hernia repair with ProFlor (Active Comparator): MRI of the pelvic area in patients who underwent inguinal hernia repair with ProFlor from 4 to 7 months before to assess tissue incorporation into the 3D scaffold
  Interventions: Device: ProFlor inguinal hernia device
- Long term post inguinal hernia repair with ProFlor (Active Comparator): MRI of the pelvic area in patients who underwent inguinal hernia repair with ProFlor after 8 months and beyond to assess tissue incorporation into the 3D scaffold
  Interventions: Device: ProFlor inguinal hernia device

INTERVENTIONS:
Device: ProFlor inguinal hernia device — Device follow up after inguinal hernia repair with ProFlor

SUMMARY:
Demonstrating through MRI sequuences the regenerative features of the 3D inguinal hernia scaffold ProFlor

DETAILED DESCRIPTION:
The biological response of the 3D inguinal hernia scaffold ProFlor has been evaluated through MRI signal intensity (SI) at three defined post-implantation stages: short, mid and long term. The SI of ProFlor has been compared to the SI of the neighbouring muscles and fat. As additional proof, histology of tissue specimens excised at the identical post-implantation stages from porcine models in the fame of a previous experimental attempt were also evaluated. The results of this experimental trial have ben already published in 2011 - ref: A new prosthetic implant for inguinal hernia repair: its features in a porcine experimental model. Artificial Organs 2011;35(8):E181-E190

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent inguinal hernia repair with the 3D inguinal hernia scaffold ProFlor

Exclusion Criteria:

* all individuals who underwent inguinal hernia repair withouth the 3D inguinal hernia scaffold ProFlor

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
tissue incorporation into ProFlor in the short term postop. | 1- 3 weeks post implantation
  evidencing the quality of the biologic response in ProFlor through signal intensity assessment collected in the T1 TSE axial sequence and measured with region-of-interest application (ROI) positioned on three different zones, respectively in muscle, fat and tissue ingrown within ProFlor
tissue incorporation into ProFlor in the mid term postop. | 4-7 months post implantation
  evidencing the quality of the biologic response in ProFlor through signal intensity assessment collected in the T1 TSE axial sequence and measured with region-of-interest application (ROI) positioned on three different zones, respectively in muscle, fat and tissue ingrown within ProFlor
tissue incorporation into ProFlor in the long term postop. | 8 months post implantation
  evidencing the quality of the biologic response in ProFlor through signal intensity assessment collected in the T1 TSE axial sequence and measured with region-of-interest application (ROI) positioned on three different zones, respectively in muscle, fat and tissue ingrown within ProFlor

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Amato, Principal Investigator — University of Cagliari
Locations (1):
- University of Palermo - Italy, Palermo, Italy

IPD SHARING:
Plan to Share IPD: Yes
upon request within
Supporting Information: Study Protocol
Time Frame: one year after study completion
Access Criteria: email contact

REFERENCES:
- [Background] Amato G, Lo Monte AI, Cassata G, Damiano G, Romano G, Bussani R. A new prosthetic implant for inguinal hernia repair: its features in a porcine experimental model. Artif Organs. 2011 Aug;35(8):E181-90. doi: 10.1111/j.1525-1594.2011.01272.x. Epub 2011 Jul 13. PMID 21752035
- [Background] Amato G, Romano G, Agrusa A, Marasa S, Cocorullo G, Gulotta G, Goetze T, Puleio R. Biologic response of inguinal hernia prosthetics: a comparative study of conventional static meshes versus 3D dynamic implants. Artif Organs. 2015 Jan;39(1):E10-23. doi: 10.1111/aor.12416. PMID 25626584
- [Background] Amato G, Romano G, Puleio R, Agrusa A, Goetze T, Gulotta E, Gordini L, Erdas E, Calo P. Neomyogenesis in 3D Dynamic Responsive Prosthesis for Inguinal Hernia Repair. Artif Organs. 2018 Dec;42(12):1216-1223. doi: 10.1111/aor.13286. Epub 2018 Oct 14. PMID 30318605
- [Background] Amato G, Agrusa A, Puleio R, Calo P, Goetze T, Romano G. Neo-nervegenesis in 3D dynamic responsive implant for inguinal hernia repair. Qualitative study. Int J Surg. 2020 Apr;76:114-119. doi: 10.1016/j.ijsu.2020.02.046. Epub 2020 Mar 10. PMID 32169570